CLINICAL TRIAL: NCT00434486
Title: An Open-Label, Randomized, 2-Period Crossover Study to Evaluate the Potential Pharmacokinetic Interaction Between Multiple Doses of Ketoconazole and a Single Dose of SKI-606 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating Drug Interaction Between Multiple Doses of Ketoconazole and a Single Dose of SKI-606
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3160A4-104
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2007-09-12 (Estimated); Status verified 2007-09

CONDITIONS: Healthy
MeSH Terms: interventions — bosutinib

INTERVENTIONS:
Drug: SKI-606

SUMMARY:
To investigate a potential pharmacokinetic interaction between SKI-606 and ketoconazole when co-administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead ECG.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-03; Study Completion 2007-03

PRIMARY OUTCOMES:
Pharmacokinetics; safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States